CLINICAL TRIAL: NCT06709196
Title: REINFORCE - Reducing Infection-related Readmissions Following Cystectomy. a Multicentre Randomised Clinical Trial Testing Superiority of Individualised Targeted Antibiotic Prophylaxis Over Empiric Prophylaxis At Ureteral Stent Removal to Reduce Infection-related Readmissions Following Cystectomy.
Brief Title: Clinical Trial Testing Whether Targeted Antibiotic Prophylaxis Can Reduce Infections After Cystectomy Compared to Empiric Prophylaxis
Acronym: REINFORCE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Maja Vejlgaard, Coordinating investigator, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-514312-27-00; 2024-514312-27-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Cystectomy; Bladder Cancer Requiring Cystectomy; Postoperative Infections; Antibiotic Prophylaxis; Ileal Conduit
Keywords: Targeted antimicrobial prophylaxis; Infection-related readmissions
MeSH Terms: interventions — Amdinocillin Pivoxil; Amoxicillin-Potassium Clavulanate Combination; Amoxicillin; Cefuroxime; Ciprofloxacin; Linezolid; Nitrofurantoin; Trimethoprim; Trimethoprim, Sulfamethoxazole Drug Combination; Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Targeted antimicrobial prophylaxis (Experimental): The participants in this arm will receive a single-day orally administered targeted antimicrobial prophylaxis on the day of ureteral stent removal based on the microbiological analysis of a postoperative urine culture.
  Interventions: Drug: Pivmecillinam; Drug: Amoxicillin clavulanic acid; Drug: Amoxicillin; Drug: Cefuroxime; Drug: Ciprofloxacin; Drug: Linezolid; Drug: Nitrofurantoin; Drug: Trimethoprim; Drug: Sulfamethoxazole trimethoprim; Drug: Fluconazole
- Empiric antimicrobial prophylaxis (Active Comparator): The participants in this arm will receive three doses of orally administered pivmecillinam 400mg morning, noon, and evening on the day of ureteral stent removal.
  Interventions: Drug: Pivmecillinam

INTERVENTIONS:
Drug: Pivmecillinam — Orally administered pivmecillinam 400mg
  Arms: Empiric antimicrobial prophylaxis
Drug: Pivmecillinam — Orally administered targeted antimicrobial prophylaxis based on a urine culture.
  Arms: Targeted antimicrobial prophylaxis
Drug: Amoxicillin clavulanic acid — Orally administered targeted antimicrobial prophylaxis based on a urine culture.
  Arms: Targeted antimicrobial prophylaxis
Drug: Amoxicillin — Orally administered targeted antimicrobial prophylaxis based on a urine culture.
  Arms: Targeted antimicrobial prophylaxis
Drug: Cefuroxime — Orally administered targeted antimicrobial prophylaxis based on a urine culture.
  Arms: Targeted antimicrobial prophylaxis
Drug: Ciprofloxacin — Orally administered targeted antimicrobial prophylaxis based on a urine culture.
  Arms: Targeted antimicrobial prophylaxis
Drug: Linezolid — Orally administered targeted antimicrobial prophylaxis based on a urine culture.
  Arms: Targeted antimicrobial prophylaxis
Drug: Nitrofurantoin — Orally administered targeted antimicrobial prophylaxis based on a urine culture.
  Arms: Targeted antimicrobial prophylaxis
Drug: Trimethoprim — Orally administered targeted antimicrobial prophylaxis based on a urine culture.
  Arms: Targeted antimicrobial prophylaxis
Drug: Sulfamethoxazole trimethoprim — Orally administered targeted antimicrobial prophylaxis based on a urine culture.
  Arms: Targeted antimicrobial prophylaxis
Drug: Fluconazole — Orally administered targeted antimicrobial prophylaxis based on a urine culture.
  Arms: Targeted antimicrobial prophylaxis

SUMMARY:
The aim of this trial is to test whether postoperative antibiotics targeted towards bacteria in the urine can reduce the risk of infection after surgical removal of the bladder (cystectomy) compared to a standardised antibiotic prophylaxis.

Participants undergoing cystectomy will be randomly assigned to postoperatively receive (A) a standardised orally administered antibiotic prophylaxis currently given at Rigshospitalet, Copenhagen or (B) a conventional orally administered antibiotic prophylaxis targeting bacteria found in the urine postoperatively.

The investigators' hypothesis is that the targeted prophylactic antibiotic strategy will reduce the number of infection-related readmissions within 90 days of surgery compared to the standardised prophylaxis.

DETAILED DESCRIPTION:
Surgical removal of the urinary bladder (cystectomy) remains one of the most complex abdominal surgeries. The procedure carries a high risk of infectious complications, and nearly one in three patients are readmitted with infection within 90 days of surgery. Due to lack of high-evidence research on prophylactic antibiotic strategies after cystectomy, the timing, duration, and type of prophylaxis varies considerably across surgical centres and nearly always encompasses a one-size-fits-all approach with an empiric antibiotic. With antibiotic stewardship gaining ground, both patients and the community at large may benefit from a more individualised targeted approach.

The investigators aim to reduce infectious complications in the postoperative course of cystectomy by conducting an investigator-initiated randomised clinical trial testing superiority of targeted antibiotic prophylaxis after cystectomy against the current standard-of-care empiric prophylaxis.

The REINFORCE trial is a multicentre, open-label, randomised, superiority trial. Cystectomy patients will be randomly assigned with a 1:1 allocation to receive one of the following orally administered antibiotic treatments on the day of ureteral stent removal: (A) Standard-of-care arm: Three doses of pivmecillinam 400mg or (B) Intervention arm: Single-day treatment of an antibiotic susceptible to the bacteria detected in a postoperative urine sample collected during index hospitalisation. If no bacteria are detected the participant will not receive antibiotics.

Patients scheduled for cystectomy will be screened for inclusion in the urological outpatient clinic at their allocated hospital. Patients who meet the inclusion and exclusion criteria will be informed of the trial and invited to participate. After informed consent, a preoperative urine culture will be collected and analysed for microbials, and two validated EORTC quality of life questionnaires will be filled out electronically.

After cystectomy during index hospitalisation, participants will deliver a postoperative urine sample, which will be analysed for bacteria and antibiotic susceptibility, and participants will be randomised into one of the two arms.

Apart from the intervention, all participants will follow the standard-of-care pre-, peri-, and postoperative treatment as per hospital guidelines. Participants will be followed for 90 days postoperatively, where complication rates and readmission rates will be collected from the Electronic Medical Records, and participants will be asked to fill out the quality of life questionnaires again.

The primary outcome is infection-related hospital readmissions within 90 days of cystectomy. We aim for an absolute risk reduction in the infection-related readmission rate of 15% (from 29% to 14%), corresponding to a number needed to treat of six patients to reduce one infection-related readmission. With a 1:1 allocation, changing block size, power of 80%, one-sided test, significance level of 0.024 accounting for alpha spending of two sequential analyses using the O'Brien-Fleming boundaries, and an anticipated dropout rate of 5%, a total of 248 participants (124 per arm) needs to be randomised.

All randomised participants will follow an intention-to-treat analysis, regardless of adherence to protocol. If some participants do not receive the allocated treatment, a per-protocol sub-analysis will be performed. The trial utilises a group sequential design to allow for the possibility of early stopping for efficacy, futility, or safety at interim analysis, which will be performed after 50% of participants have been followed for 90 postoperative days.

International guidelines are currently unable to make evidence-based recommendations on how to avoid infections after cystectomy and current antibiotic prophylactic strategies vary greatly across centres. By performing a large multicentre randomised trial to test targeted antibiotic prophylaxis, the investigators aim to improve recovery for patients who have undergone cystectomy by reducing the risk of infections in the months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age at surgery ≥ 18 years
* Ability to understand and sign an informed consent
* Malignant or benign indication for undergoing cystectomy
* Planned ileal conduit as urinary diversion

Exclusion Criteria:

* Previous severe allergic reaction to antimicrobial treatment
* Long-term prophylactic antibiotic treatment which is expected to be continued after the cystectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Infection-related readmission rate | 90 days after surgery
  The rate of readmissions where the main cause of readmission is symptoms of infection.

SECONDARY OUTCOMES:
Postoperative complications | 30 and 90 days after surgery
  Postoperative complications using the validated Clavien-Dindo classification score, ranging from 1-5 where 1-2 are minor complications and 3-5 are major complications.
Postoperative readmissions | 30 and 90 days after surgery
  All-cause postoperative readmissions, including the the main cause, timing, and duration.
Days alive and out of hospital | 30 and 90 days after surgery
  The number of days that the participants are alive and not admitted to the hospital.
Quality of life | 90 days after surgery
  Quality-of-life using the validated European Organisation of Research and Treatment of Cancer (EORTC) Quality of Life Core Questionnaire (QLQ-C30). Results will be presented as scores ranging from 0-100 where high scores in the global health status and functional scales represent a better quality of life and high scores in the symptom scales represent a high level of symptomatology.
Quality of life | 90 days after surgery
  Quality-of-life using the validated European Organisation of Research and Treatment of Cancer (EORTC) Quality of Life Muscle-invasive Bladder Cancer Questionnaire (QLQ-BLM30). Results will be presented as scores ranging from 0-100 where high scores in the global health status and functional scales represent a better quality of life and high scores in the symptom scales represent a high level of symptomatology.
Microbiological findings | 90 days after surgery
  Microbiological findings and antimicrobial susceptibility analyses in pre- and postoperative microbiological samples.
Antimicrobial treatment | 90 days after surgery
  All antimicrobial treatment registered in the Electronic Medical Records.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Røder, Prof, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (5):
- Denmark (5):
  - Department of Urology, Aalborg University Hospital, Aalborg
  - Department of Urology, Aarhus University Hospital, Aarhus
  - Department of Urology, Rigshospitalet, Copenhagen
  - Department of Urology, Herlev and Gentofte Hospital, Herlev
  - Department of Urology, Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vejlgaard M, Stroomberg HV, Ynddal MS, Moser C, Joensen UN, Roder A. Multicentre, open-label, phase IV, randomised trial testing superiority of individualised targeted antibiotic prophylaxis over empiric prophylaxis at ureteral stent removal following cystectomy: study protocol for the REINFORCE trial. Trials. 2025 Jul 28;26(1):258. doi: 10.1186/s13063-025-08981-w. PMID 40722189